CLINICAL TRIAL: NCT02849834
Title: Study of Sensory-motor Cortex Plasticity After Motor Cortex Stimulation in Healthy Subject and Chronic Pain Patients
Brief Title: Cortical Plasticity After Motor Cortex Stimulation in Healthy Subject and Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2008-505; 2008-A01437-38 (Other: ID-RCB)
Record Dates: First submitted 2016-07-26; First posted 2016-07-29 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Stimulation of the Motor Cortex (SCM); Pharmacoresistant; rTMS
MeSH Terms: conditions — Neuralgia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- healthy volunteers (Active Comparator)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Patients with resistant pain (Experimental)
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — 20Hz and Theta Burst stimulation, both at 80% of motor threshold in contralateral intrinsic hand muscles. Five consecutive days of each mode of stimulation, separated by a minimum of 4 weeks. Daily self-monitoring of pain, sleep quality and fatigue by mans of a 10-item questionnaire

SUMMARY:
The primary aim of this study is to evaluate the induction of sensory-motor cortex plasticity after motor cortex stimulation in healthy subjects, using laser-evoked nociceptive cortical potentials, and in chronic neuropathic pain patients using functional MRI. As a secondary goal, the project will analyse possible correlations between the magnitude of cortical plasticity and that of the pain-relieving effect.

In healthy subjects, cortical plasticity is evaluated by the comparison of somatosensory cortical maps before and after two isolated sessions of 20 Hz and theta-burst rTMS, in a cross-over randomized study.

Two sessions of 5 consecutive days of rTMS are proposed to the patients with a minimum of 4 weeks between the two sessions, defined by 20 Hz and theta-burst stimulation in a cross-over randomized order. Cortical plasticity of the motor cortex is evaluated via functional MRI (motor activation) performed before the first rTMS session and the last day of each session of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects aged from 18 to 70 years, male or female, with social protection, fully informed and having given their written consent.
* patients :

  * aged from 18 to 80 years, male or female, with social protection , fully informed and having given their written consent.
  * unilateral pharmacoresistant neuropathic pain during at least one year,
  * without any change of the pharmacological treatment since at least one month

Exclusion Criteria:

* for healthy subjects only:
* history of chronic pain
* analgesic medication within 24h before stimulation

For patients only: new analgesic treatment within 1 month before consent

for both:

* drug addiction, headache, epilepsy history
* ferromagnetic intracranial device
* implanted stimulator
* absence of contraceptive method for women of childbearing age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-11; Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
cortical plasticity induced by rTMS - - Somatosensory evoked potentials | just before the isolated 20 Hz or theta-burst stimulation for healthy subjects
  Assessment of plastic changes induced in sensori-motor cortex by the application of repetitive magnetic stimulation in healthy subjects and chronic pain patients.
  * In healthy subjects, mapping of cortical responses amplitude and source reconstruction techniques (dipole modelisation, BESA) before / after a single rTMS session
  * In chronic pain patients, contrast analysis between extent and location of motor activations (to hand, foot and mouth contraction) before / after one week of daily rTMS, analysed with Statistical Parametric Mapping (SPM12)
cortical plasticity induced by rTMS - - Somatosensory evoked potentials | just after the isolated 20 Hz or theta-burst stimulation for healthy subjects
  Assessment of plastic changes induced in sensori-motor cortex by the application of repetitive magnetic stimulation in healthy subjects and chronic pain patients.
  * In healthy subjects, mapping of cortical responses amplitude and source reconstruction techniques (dipole modelisation, BESA) before / after a single rTMS session
  * In chronic pain patients, contrast analysis between extent and location of motor activations (to hand, foot and mouth contraction) before / after one week of daily rTMS, analysed with Statistical Parametric Mapping (SPM12)
cortical plasticity induced by rTMS -- fMRI | within 1 week before the first day of stimulation (20 Hz or theta-burst) for the patients
  Assessment of plastic changes induced in sensori-motor cortex by the application of repetitive magnetic stimulation in healthy subjects and chronic pain patients.
  * In healthy subjects, mapping of cortical responses amplitude and source reconstruction techniques (dipole modelisation, BESA) before / after a single rTMS session
  * In chronic pain patients, contrast analysis between extent and location of motor activations (to hand, foot and mouth contraction) before / after one week of daily rTMS, analysed with Statistical Parametric Mapping (SPM12)
cortical plasticity induced by rTMS -- fMRI | after the 5th day of stimulation (20 Hz or theta-burst) for the patients
  Assessment of plastic changes induced in sensori-motor cortex by the application of repetitive magnetic stimulation in healthy subjects and chronic pain patients.
  * In healthy subjects, mapping of cortical responses amplitude and source reconstruction techniques (dipole modelisation, BESA) before / after a single rTMS session
  * In chronic pain patients, contrast analysis between extent and location of motor activations (to hand, foot and mouth contraction) before / after one week of daily rTMS, analysed with Statistical Parametric Mapping (SPM12)

SECONDARY OUTCOMES:
Nonparametric (Chi-2) contrast of dichotomized pain reports before/after rTMS and extent of fMRI activation change (also dichotomized) MRI T1 3D and T2* | within 1 week before the first day of stimulation Stats after 40 patients studied.
Nonparametric (Chi-2) contrast of dichotomized pain reports before/after rTMS and extent of fMRI activation change (also dichotomized) MRI T1 3D and T2* | after the 5th day of stimulation. Stats after 40 patients studied.
Linear and nonlinear correlation between the magnitude of induced cortical plasticity and the magnitude of pain relief induced by rTMS. MRI T1 3D and T2*, | within 1 week before the first day of stimulation Stats after 40 patients studied.
Linear and nonlinear correlation between the magnitude of induced cortical plasticity and the magnitude of pain relief induced by rTMS. MRI T1 3D and T2*, | after the 5th day of stimulation. Stats after 40 patients studied.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie ANDRE-OBADIA, MD, Principal Investigator — Service d'Exploration, Centre Hospitalier Lyon Est, Hospices civils de Lyon, Lyon, F-69495, France et NeuroPain lab - CRNL (Inserm U1028 - UCBL)
Locations (1):
- Service d'Exploration, Centre Hospitalier Lyon Est, Hospices civils de Lyon, Lyon, F-69495, France et NeuroPain lab - CRNL (Inserm U1028 - UCBL), Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andre-Obadia N, Hodaj H, Hodaj E, Simon E, Delon-Martin C, Garcia-Larrea L. Better Fields or Currents? A Head-to-Head Comparison of Transcranial Magnetic (rTMS) Versus Direct Current Stimulation (tDCS) for Neuropathic Pain. Neurotherapeutics. 2023 Jan;20(1):207-219. doi: 10.1007/s13311-022-01303-x. Epub 2022 Oct 20. PMID 36266501